CLINICAL TRIAL: NCT00477360
Title: Humeral Resurfacing Hemiarthroplasty. Phase 2: Prospective Cohort Study
Brief Title: Humeral Resurfacing Hemiarthroplasty
Acronym: CAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Calgary (Other)
Collaborators: DePuy International (Industry); Johnson & Johnson (Industry)
Responsible Party: Dr. Richard Boorman, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 15052007
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Advanced Glenohumeral Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): C.A.P
  Interventions: Device: Humeral surface replacement hemiarthroplasty (CAP)

INTERVENTIONS:
Device: Humeral surface replacement hemiarthroplasty (CAP) — C.A.P hemiarthroplasty

SUMMARY:
The primary objective of this study is to examine quality of life outcomes in patients who have undergone a humeral surface replacement hemiarthroplasty.

DETAILED DESCRIPTION:
Resurfacing arthroplasty is gaining popularity for the reconstruction of advanced shoulder arthritis. New generation re-surfacing prostheses are engineered to anatomically restore a smooth articulating surface to the humeral head, while preserving bone stock, and potentially minimizing the risk for diaphyseal fracture. The results for shoulder resurfacing prostheses have largely been reported in retrospective reviews and have been very favorable. The purpose of this multi-centered, prospective study will be to determine the extent to which patient self-assessed outcomes (American Shoulder and Elbow Society (ASES) Score) following humeral resurfacing improve compared to pre-operative ASES scores.

ELIGIBILITY:
Pre-Operative Inclusion Criteria:

* Failed standard non-surgical management (analgesics, nsaids, physiotherapy, activity modification)
* Persistent pain and disability for at least 6 months
* Imaging demonstrates advanced humeral head cartilage loss

Pre-Operative Exclusion Criteria:

* Active or systemic joint infection
* Significant muscle paralysis of shoulder girdle
* Charcot's Arthropathy
* Major medical illness (life expectancy <2years)
* Unable to speak and read English/French
* Psychiatric illness that precludes informed consent
* Unwilling/unable to remain in study for one year

Intra-Operative Inclusion Criteria:

Advanced humeral head cartilage loss AND ONE of:

* minimal/no glenoid cartilage loss
* complete glenoid cartilage loss and no bony erosion
* complete glenoid cartilage loss and concentric bony erosion with no humeral anterior/posterior subluxation

Intra-Operative Exclusion Criteria:

* Eccentric glenoid erosion with biconcavity of glenoid and subluxation of humeral head
* Inability of humeral head to support the CAP surface replacement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
American Shoulder And Elbow Surgeons Shoulder Index (ASES) | 24 months post-operative

SECONDARY OUTCOMES:
Constant Score | 24 months post-operative
Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | 24 months post-operative
Simple Shoulder Test (SST) | 24 months post-operative
Radiographic Evaluation | 3 months + yearly post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Richard Boorman, Principal Investigator — University of Calgary; Dr. Dianne Bryant, Principal Investigator — Western University, Canada
Locations (1):
- University of Calgary Sport Medicine Centre, Calgary, Alberta, Canada